CLINICAL TRIAL: NCT05587621
Title: "Intensive Lipid-Lowering Therapy Guided by a Cloud-based Software System (CLIMEDO GmbH) in Patients With ST-Elevation and Non-ST-Elevation Myocardial Infarctions" (Germany on Target)
Brief Title: Intensive Lipid-lowering in Patients With STEMI and NSTEMI (Germany on Target)
Acronym: GoT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5219-07/17
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-09

CONDITIONS: ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction; LDL-cholesterol
Keywords: STEMI, NSTEMI; LDL-C; target attainment
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; evolocumab; alirocumab; ALN-PCS; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: randomized trial to compare a cloud-based software system with standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cloud-based software (Active Comparator): cloud-based software system (CLIMEDO GmbH) will support patients in ESC/EAS LDL-C target attainment (< 55mg/dl/1.4 mol/L)
  Interventions: Drug: statins, ezetimibe, bempedoic acid, evolocumab, alirocumab, inclisiran
- Standard Care (Placebo Comparator): Patients will be treated by general practitioners (GPs) after hospital discharge. The discharge letter will recommend ESC/EAS dyslipidemia LDL-cholesterol targets (< 55mg/dl/1.4 mol/L)
  Interventions: Drug: statins, ezetimibe, bempedoic acid, evolocumab, alirocumab, inclisiran

INTERVENTIONS:
Drug: statins, ezetimibe, bempedoic acid, evolocumab, alirocumab, inclisiran — dietary advice for low cholesterol food
  Other Names: dietary advice

SUMMARY:
Intensive Lipid-Lowering Therapy guided by a cloud-based Software System (CLIMEDO GmbH) improves (European Society of Cardiolofgy/European Atherosclerosis Society) ESC/EAS-guideline recommended LDL-cholesterol target attainment and adherence in patients with ST-Elevation Myocardial (STEMI) and Non-ST-Elevation Myocardial Infarctions (NSTEMI).

DETAILED DESCRIPTION:
Patients admitted to the Jena University Hospital (UKS) and 9 other University hospitals in Germany with an ST-elevation or Non-ST-elevation myocardial infarction (STEMI) will be randomized to standard care or a software-based tool (CLIMEDO GmbH) to monitor low-density cholesterol (LDL-C) levels and close follow-ups to achieve ESC/EAS-guideline recommended LDL-C goals.

In this multi-center, prospective, randomized, interventional trial we propose that using a cloud-based software system (CLIMEDO GmbH) is superior to standard care in terms of LDL-C target attainment at 6 months and adherence over a time period of 12 months.

In the software group LDL-C levels will be monitored on admission, after 1,6, 12, 16, 20 weeks and after 6, 12 and 24 months. In the standard care group patients' LDL-C levels will be determined on admission after 6, 12 and 24 months. The primary endpoint is LDL-C target attainment at 6 months in both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with ST- and Non-ST-elevation myocardial infarctions

Exclusion Criteria:

* patient without informed concent
* patients in cardiogenic shock
* patients with contraindication to lipid-lowering therapy
* patients on lipid-lowering medications on admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
LDL-C | 6 months
  LDL-C target attainment (ESC/EAS dyslipidemia guidelines)

SECONDARY OUTCOMES:
side-effects of lipid lowering therapy | 6 months
  muscle pain, hair loss, dizziness, joint pain, depression
adherence to LLT | 12 months
  regular LLT

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Weingärtner, MD, Principal Investigator — Jena University Hospital
Locations (10):
- Germany (10):
  - University Hospital Jena, Jena, Thuringia
  - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No